CLINICAL TRIAL: NCT02086214
Title: Pressure Therapy in the Treatment of Upper Arm of Cerebral Palsy Children
Acronym: PROPENSIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Marc Sautelet Centre (Villeneuve d'Ascq, France) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011_01; N°19/16, Axe 1.11, (Other Grant/Funding Number: PHRC-2011); 2011-A01129-32 (Other: ID-RCB number, AFSSAPS)
Record Dates: First submitted 2014-02-17; First posted 2014-03-13 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy
Keywords: Upper limb; Proprioceptive pressure therapy; Children; Assisting Hand Assessment performance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proprioceptive pressure therapy (Experimental): Proprioceptive pressure therapy using a a LYCRA® compressive sleeve initially used in burn therapy : 15 to 25 mmHg.
  Interventions: Device: Proprioceptive pressure therapy
- Control (Placebo Comparator): LYCRA® non-compressive sleeve initially used in burn therapy : < 5 mmHg.
  Interventions: Device: Control

INTERVENTIONS:
Device: Proprioceptive pressure therapy — Proprioceptive pressure therapy using a a LYCRA® compressive sleeve initially used in burn therapy : 15 to 25 mmHg.
  Other Names: Proprioceptive pressure therapy by Medical Z
  Arms: Proprioceptive pressure therapy
Device: Control — LYCRA® non-compressive sleeve initially used in burn therapy : < 5 mmHg.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the efficacy of a 6 months upper arm proprioceptive pressure therapy on Assisting Hand Assessment ("AHA") performance in Cerebral Palsy (CP). To perform this study, 80 CP patients aged of 5 to 10 years old will be included in a multicentric, double blind, prospective parallel-group randomized study. Treatment will be a pressure therapy using a LYCRA® compressive sleeve initially used in burn therapy. Primary outcome is to increase of 60% of AHA performance. The secondary outcome are to increase Quality of Upper Extremity Skill Test (QUEST), quality of life and improve Somatosensory Evoked Potentials (SEP).

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of a 6 months upper arm proprioceptive pressure therapy on Assisting Hand Assessment ("AHA") performance in Cerebral Palsy (CP). To perform this study, 80 CP patients aged of 5 to 10 years old will be included in a multicentric, double blind, prospective parallel-group randomized study. Treatment will be a pressure therapy using a LYCRA® compressive sleeve initially used in burn therapy. Primary outcome is to increase of 60% of AHA performance. The secondary outcome are to increase Quality of Upper Extremity Skill Test (QUEST), quality of life and improve Somatosensory Evoked Potentials (SEP)

ELIGIBILITY:
Inclusion Criteria:

* Children with upper limb with pre/peri birth etiologic CP.
* Children aged 5 to 10 years

Exclusion Criteria:

* Children with language dysfunction
* LYCRA® allergia
* Botulic Toxin injection on upper limb 4 month before inclusion

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment performance | 6 months
  Assisting Hand Assessment performance is a functional test to assess hand function for children with unilateral upper limb disabilities.

SECONDARY OUTCOMES:
Upper Extremity skill Test (QUEST) | 6 months
  Upper Extremity skill Test is a functional test to assess upper limb mobility for children with unilateral upper limb disabilities.
Somatosensory Evoked Potentials (SEP) | 6 months
  Somatosensory Evoked Potentials (SEP) is a functional test to assess sensory nerve conduction

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GOTTRAND, MD, Principal Investigator — Centre Marc Sautelet, Villeneuve d'Ascq, France
Locations (5):
- France (5):
  - CHU, Amiens
  - Service d'Education et de Soins Spécialisés à domicile_APF de Creil, Creil
  - CHU, Reims
  - Centre de Soins de Suite et de Réadaptation Pédiatrique Spécialisé_Centre Paul Dottin, Toulouse
  - Centre Marc Sautelet, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gerard A, Toussaint-Thorin M, Mohammad Y, Letellier G, Fritot S, Masson S, Duhamel A, Donskoff C, Zagame Y, Beghin L, Gottrand L. PROPENSIX: pressure garment therapy using compressive dynamic Lycra(R) sleeve to improve bi-manual performance in unilateral cerebral palsy: a multicenter randomized controlled trial protocol. Trials. 2022 Feb 5;23(1):117. doi: 10.1186/s13063-022-06041-1. PMID 35123557